CLINICAL TRIAL: NCT04733430
Title: Landsteiner Lung Cancer Research Platform (LALUCA) A Prospective Analysis of Lung Cancer Diagnosis and Management in Clinical Practice
Brief Title: LALUCA Research Platform A Prospective Analysis of Lung Cancer Diagnosis and Management in Clinical Practice
Acronym: LALUCA
Status: Recruiting | Type: Observational
Sponsor: Karl Landsteiner Institute for Lung Research and Pneumological Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: LALUCA Project Plan Version 5
Record Dates: First submitted 2021-01-18; First posted 2021-02-02 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: NGS Testing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective analysis of the diagnosis and treatment of lung cancer in a real-world setting. The aim of the project is to establish a clinical platform to collect representative data on molecular testing, sequence of systemic tumor therapy and other therapies, and disease progression of patients with lung cancer. A special focus will be on molecular biomarker testing and reflex NGS testing. Another aim of the registry is the collection of quality indicators in lung cancer care. The results of the register will be used to describe the current state of care and to develop it further for the future.

DETAILED DESCRIPTION:
The identification of driver-mutations, whose gene product can be specifically inhibited by targeted therapies, has markedly changed the diagnostic and therapeutic landscape for this tumor entity, leading to improved outcomes for patients with metastatic NSCLC.

The use of next generation sequencing (NGS) allows for detection of a multitude of different druggable mutations. In absence of a curative treatment approach and a druggable mutation the prognosis of lung cancer remains poor.

Thorough knowledge of the treatment reality, e.g. characteristics, diagnostic, treatment and outcome of unselected patients in real-Iife practice, is crucial to evaluate and improve the quality of care for patients with lung cancer.

The purpose of this project is to set up a clinical platform to document representative data on molecular testing, sequence of systemic treatment and other treatment modalities, and course of disease in patients with lung cancer. A particular focus is on molecular biomarker testing and NGS of patients before the start of first-line treatment. The data shall be used to assess the current state of care and to develop recommendations concerning topics that can be improved.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically confirmed lung cancer
* Age ≥ 18 years
* Able to understand and willing to sign written Informed Consent and to complete patient-reported-outcome assessment instruments

Exclusion Criteria:

-

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All unselected patients diagnosed with lung cancer at the research sites. The study is intended to commence at two sites in Vienna, with subsequent invitation of participation of other sites.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
NGS Testing | through study completion, an average of 5 years
  To assess molecular biomarker testing and indicators of the quality of care in patients with lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Georg-Christian Funk, MD, Principal Investigator — 2nd Medical Department with Pneumology
Locations (1):
- Karl Landsteiner Institut für Lungenforschung und Pneumologische Onkologie, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No